CLINICAL TRIAL: NCT02591537
Title: Prospective, Randomized, Single Center, Controlled Evaluation of the Effectiveness of OxyGenesys Topical Dissolved Oxygen Dressing in Accelerating the Healing of Split Thickness Skin Graft Donor Sites Using the NWU Abdominoplasty Scar Model
Brief Title: OxyGenesys Dissolved Oxygen Dressing; Abdominoplasty at Northwestern University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halyard Health (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100-15-0001
Record Dates: First submitted 2015-10-12; First posted 2015-10-29 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-08

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OxyGenesys Dissolved Oxygen Dressing (Experimental): OxyGenesys Dissolved Oxygen Dressing will be applied.
  Interventions: Device: OxyGenesys Dissolved Oxygen Dressing
- Standard Tegaderm Dressing (No Intervention): Tegaderm will be applied.

INTERVENTIONS:
Device: OxyGenesys Dissolved Oxygen Dressing — 1/2 of the abdominal wounds will be covered with Oxygenesys Dissolved Dressing.
  Arms: OxyGenesys Dissolved Oxygen Dressing

SUMMARY:
Twelve acute wounds (6 on either side of the umbilicus) will be surgically created in the lower abdominal area. One side of the umbilicus will be randomized to Oxygenesys treatment arm and the other side will be receiving a standard Tegaderm treatment arm. Time to wound healing will be observed over 14 days.

DETAILED DESCRIPTION:
At least 12 study visits will occur over a 3 month timeframe. Twelve acute wounds (6 on either side of the umbilicus) will be surgically created in the lower abdominal area. One side of the umbilicus will be randomized to Oxygenesys treatment arm and the other side will be receiving a standard Tegaderm treatment arm. Time to wound healing will be observed over 14 days (follow up assessments include wound photography, pain scores, wound biopsies, exudate collection, gene expression and proteomic analysis, scar assessment and adverse event collections. Study visits will occur at:

Prescreening Visit; Day of wounding; Day 2; Day 7; Day 8-14 (until all wounds have healed); Day 28; Day 42; Abdominoplasty Surgery. An abdominoplasty will occur after day 42.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females aged 21-85 years. Female subjects of child bearing potential must be using method(s) of contraception acceptable to the Investigator and agree to do so from at least the screening visit until one month after administration of the final study dressing.
* Subject is willing to undergo the creation of twelve experimental donor sites 1.0" x 1.0" in size with a depth between 0.0012"-0.0018" taken from the abdomen per a modification of the Northwestern Abdominoplasty Scar Model
* Subjects who are medically acceptable candidates for abdominoplasty (BMI approximately 25-35 kg/m2) as determined by per-study laboratory assessment and clinical evaluation.
* Willingness to provide informed consent and to comply with the requirements of this protocol for the full duration of the study.

Exclusion Criteria:

* Subjects who have received treatment with systemic steroids during the 30 days prior to study enrollment.
* Subjects who have received immunosuppressive drugs, radiation or chemotherapy during the three months prior to study enrollment.
* Subjects with a history of malignancy in the previous three years.
* Subjects with uncontrolled diabetes (A1C > 8%).
* Subjects who are current smokers or have any significant pack-year history of smoking (>1 pack-year).
* Subjects with diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerability or efficacy.
* Subjects who have previously had skin grafts harvested from the area to be studied.
* Subjects with a skin disorder (other than chronic venous ulcers) that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Subjects with extensive severe striae that would make it difficult to perform a skin graft on the abdomen and/or evaluate the final scar appearance.
* Subjects with a history of clinical significant hypersensitivity to any of the surgical dressings to be used in this trial.
* Subjects who are taking, or have taken any Investigational drugs within 3 months prior to the screening visit.
* Subjects who are participating in other research Investigations.
* Subjects requiring treatment with medications(s) that are known to interfere with wound healing.
* Subjects who are or who become pregnant up to and including Day 0 or who are lactating.
* Subjects who, in the opinion of the Investigator, are not likely to complete the trial for whatever reason, including significant comorbidities that may adversely affect survival or ability to attend follow up visits.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant was assigned to both study groups (acted as her own control), as four wounds on one side of each participant were treated with OxyGenesys dressing, and four wounds on the opposite side of each participant were treated with the Tegaderm control dressing.
Units Other Than Participants: wounds
Groups:
- Standard Tegaderm Dressing: Standard Tegaderm Dressing will be applied.
Period: Overall Study
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Started | 8; 32 wounds | 8; 32 wounds
Completed | 8; 32 wounds | 8; 32 wounds
Not Completed | 0; 0 wounds | 0; 0 wounds

BASELINE CHARACTERISTICS:
Population: Each participant was assigned to both study groups (acted as her own control), as four wounds on one side of each participant were treated with OxyGenesys dressing, and four wounds on the opposite side of each participant were treated with the Tegaderm control dressing. In some instances, not all of the participants contributed data to outcomes.
Units Other Than Participants: wounds
Groups:
- Total: Total of all reporting groups
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing | Total
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (wounds) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12) | 41.6 (12) | 41.6 (12)
Sex: Female, Male [Count of Units; unit: wounds]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Units; unit: wounds]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: wounds]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Healing in Days.
Description: Wound healing will be defined as 90% re-epithelialization. Mean time to healing will be compared between the OxyGenesys treated sites and the control treated sites.
Time Frame: 14 days
Population: Each participant was assigned to both study groups (acted as her own control), as four wounds on one side of each participant were treated with OxyGenesys dressing, and four wounds on the opposite side of each participant were treated with the Tegaderm control dressing.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: wounds
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 8 | 8
Number analyzed (wounds) | 32 | 32
days | 13.1 (2.8) | 12.5 (2.1)

2. Secondary Outcome: Wound Degree of Epithelialization Percent Change by Digital Photography at Each Time Point Post Wounding.
Description: Wound degree of epithelialization percent change by digital photography at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of epithelialization
Units Other Than Participants: wounds
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 8 | 8
Number analyzed (wounds) | 32 | 32
percentage of epithelialization | 81.4 (15.7) | 91.3 (8.3)

3. Secondary Outcome: Pain on Test Versus Control Side Using a Wong-Baker Scale.
Description: Subjects will report pain level on each side of their abdomen at day 14. The Wong-Baker scale is: 0 points = no hurt, 2 = hurts little bit, 4 = hurts little more, 6 = hurts even more, 8 = hurts whole lot, 10 = hurts worst. A grand mean and standard deviation (reported below) were determined by combining participant scores.The identical group mean and standard deviation values reported below are correct.
Time Frame: Day 14
Population: Each participant was assigned to both study groups (acted as her own control), as four wounds on one side of each participant were treated with OxyGenesys dressing, and four wounds on the opposite side of each participant were treated with the Tegaderm control dressing. Five participants did not report their day 14 measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wounds
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 3 | 3
Number analyzed (wounds) | 12 | 12
units on a scale | 0.7 (1.2) | 0.7 (1.2)

4. Secondary Outcome: Biopsy & Histology of Wounds.
Description: Biopsies will be taken from all wounds at day 28. Analysis of tissue samples will specifically evaluate differences and rates of collagen deposition, angiogenesis and re-epithelialization between the two study arms.
Time Frame: Day 28
Population: Each participant was assigned to both study groups (acted as her own control). Samples were collected, but not analyzed because the comparative broad healing endpoints did not provide compelling evidence for tissue processing. No data are presented because the Outcome Measure has zero total participants analyzed.
Units Other Than Participants: wound biopsies
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 0 | 0
Number analyzed (wound biopsies) | 0 | 0

5. Secondary Outcome: Scar Quality Analysis; Modified Vancouver Scar Scale (MVS)
Description: Scar quality will be assessed and analyzed between the two groups using the Modified Vancouver Scar Scale at day 42. The MVS assessment is the tool that the Investigator will use to evaluate scar pliability (0 points = normal, 1 = supple, 2 = yielding, 3 = firm, 4 = adherent), height (0 = normal, 1 = 1-2 mm, 2 = 3-4 mm, 3 = 5-6 mm, 4 = > 6 mm), vascularity (0 = normal, 1 = pink, 2 = red, 3 = purple), and pigmentation (0 = normal, 1 = slight, 2 = moderately, 3 = severely). An average score for each participant was calculated by combining scores from each subscale. Average participant scores in each study group were combined to produce a grand mean and standard deviation for each group (reported below).
Time Frame: Day 42
Population: Each participant was assigned to both study groups (acted as her own control), as four wounds on one side of each participant were treated with OxyGenesys dressing, and four wounds on the opposite side of each participant were treated with the Tegaderm control dressing. One participant did not report for her day 42 measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wounds
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 7 | 7
Number analyzed (wounds) | 28 | 28
units on a scale | 3.8 (1.7) | 3.8 (1.4)

6. Secondary Outcome: Scar Quality Analysis; Visual Analogue Scale
Description: Scar quality of each study participant was assessed by using the Visual Analogue Scale (VAS) at day 42. The VAS is an 11-point scale that ranges from 0 (normal skin) to 10 (worst possible scar). The values on the scale indicate the observer's global impression of the scar (lower numbers are better than higher numbers).
Time Frame: Day 42
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wounds
Groups:
- Standard Tegaderm Dressing: Standard Tegaderm Dresssing will be applied.
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 7 | 7
Number analyzed (wounds) | 28 | 28
units on a scale | 5.8 (2) | 5.9 (2.2)

7. Secondary Outcome: Scar Quality Analysis; Elastometer
Description: Scar quality was to be assessed for each study participant using an elastometer at day 42. An elastometer is used to assess scar elasticity. Unfortunately, the data for this study endpoint were not collected properly, and despite our best efforts, there is no way to resolve this issue. Thus, no data can be reported for this study outcome.
Time Frame: Day 42
Population: Data were not collected.
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Scar Quality Analysis; Colorimeter
Description: Scar quality was to be assessed for each study participant using a colorimeter at day 42. A colorimeter was to be used to measure the extent of erythema, and melanin content, of the skin. Unfortunately, the data for this study endpoint were not collected properly, and despite our best efforts, there is no way to resolve this issue. Thus, no data can be reported for this study outcome.
Time Frame: Day 42
Population: Data were not collected.
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Tegaderm Dressing
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OxyGenesys Dissolved Oxygen Dressing (N=8) | Standard Tegaderm Dressing (N=8)
folliculitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No